CLINICAL TRIAL: NCT05165862
Title: Evaluation and Monitoring of the Protocol for the Management of Post Operative Atrial Fibrillation Based on Intravenous Beta-blockers in Cardiac Surgery
Brief Title: Evaluation and Monitoring of the Protocol Post Operative Atrial Fibrillation
Acronym: ETOFIB
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: ETOFIB (29BRC20.0038)
Record Dates: First submitted 2020-09-24; First posted 2021-12-21 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Post Operative Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Objectives The aims of this study is to evaluate the efficacy and tolerance of our post-operative AF management protocol after cardiac surgery, including beta-blockers, digoxin, amiodarone.

Methods This study concerns patients From brest university Hospital who underwent cardiac surgery between November 2019 and November 2021. Patients with a previous history of atrial arrhythmias were excluded. The primary endpoint is assess effectiveness of service protocol to maintain cardiac frequency below. 110 bpm. The secondary endpoints included hemodynamic tolerance and outcomes.

DETAILED DESCRIPTION:
Background Atrial fibrillation (AF) is the most common complication after open heart surgery. Its reported incidence is about 30%, and it is associated with a significant increase rate of thromboembolic events, respiratory failure, a longer lenght of stay in hospital and mortality. (1 ;2) Gillinov's study has shown equivalent effectiveness of a rhythm control and rate control strategy, in AF patients after cardiac surgery, with increased side effects in patients treated with rhythm control agents. (3) The introduction of beta-blockers can be poorly tolerated hemodynamically in patients hospitalized in intensive care unit, unless untroducing a cardio-selective beta-blocker..

Methods Patients who underwent a cardiac surgery from Novembre 2019 to Novembre 2021 were included. Patients with a previous history of atrial arrhythmias were excluded. The primary endpoint is assess effectiveness of service protocol to maintain cardiac frequency below. 110 bpm. The secondary endpoints included hemodynamic tolerance and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* POAF after cardiac surgery non-opposition formulated

Exclusion Criteria:

* pregnant woman opposition hemodynamic unstability with inotropic drugs or CI<2 L/min/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: POAF after cardiac surgery, hospitalized in ICU
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-10-16 (Actual); Study Completion 2021-10-16 (Actual)

PRIMARY OUTCOMES:
Heart Rate | 72 hours (3 days)
  HR < 110 BPM

SECONDARY OUTCOMES:
sinusal Rythm | 72hours ( 3 days)
  time to be back in sinusal rythm

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest - Service d'anesthésie-Réanimation, Brest, France